CLINICAL TRIAL: NCT02784691
Title: Efficiency and Usability of the Iontophoretic Patch Feeligreen Diclofenac in Treating Acute Osteoarthritic Knee Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of logistical problems
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-PP-15
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental)
  Interventions: Device: Feeligreen patch

INTERVENTIONS:
Device: Feeligreen patch

SUMMARY:
The aim of the study is to evaluate the antalgic efficacity of Feeligreen® patch on osteoarthritic knee pain acute. This patch work by diffusion controlled by iontophoresis allowing an improvement of transdermal diffusion of active (Diclofenac).

ELIGIBILITY:
Inclusion Criteria:

* Patients with age above 70 years,
* Having a knee Arthritis (unilateral or bilateral) for at least 6 months,
* Pain intensity ≥ 40 mm on a visual analog scale (VAS)
* Lack of analgesic treatment or analgesic,

Exclusion Criteria:

* Cognitive disorders : moderate to severe stage or not allowing an understanding of the VAS (as determined by the clinician)
* A history of chronic inflammatory rheumatic disease,
* Diagnosis of osteoarthritis of secondary origin,
* Non-steroidal anti-inflammatory medication within 7 days prior to inclusion,
* Diagnosis of severe hepatic and renal insufficiency, gastrointestinal bleeding, severe heart failure,
* Allergy to diclofenac or similar activity substances such as other NSAIDs, aspirin, excipients,
* Damaged skin

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Intensity reduction of pain | 2 days
  Measured by Visual Analog Scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No